CLINICAL TRIAL: NCT00906958
Title: Comparison of the Efficacy and Subjective Comfort of a Modified AutoSet Device With an Existing AutoSet Device (VPAP Auto) in Treating Obstructive Sleep Apnea
Brief Title: Modified AutoSet Device vs Existing AutoSet Device, the Assessment of Efficacy and Subjective Comfort of the Treatment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08177-0608; NCT00773396 (obsolete NCT alias)
Record Dates: First submitted 2009-05-13; First posted 2009-05-21 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Nexus Flow Generator (Experimental): Participants were randomised to Nexus Flow Generator group for one night.
  Interventions: Device: Nexus Flow Generator
- VPAP Flow Generator 25 (Active Comparator): Participants were randomised to VPAP Flow Generator 25 group for one night.
  Interventions: Device: VPAP Flow Generator 25

INTERVENTIONS:
Device: Nexus Flow Generator — The modified device to be assessed in this study will act in a similar way to the existing device, VPAP Auto, but utilises an improved algorithm which should maintain or enhance the effectiveness of the treatment.
  Arms: Nexus Flow Generator
Device: VPAP Flow Generator 25 — Exiting VPAP Auto 25 Flow Generator with A10 Algorithm
  Arms: VPAP Flow Generator 25

SUMMARY:
The purpose of this study is to determine if the performance of the modified AutoSet device is equivalent or better than the existing AutoSet device (VPAP Auto) in the efficacy of the treatment and the subjective comfort.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterised by a partial or complete collapse of the upper airway during sleep. The treatment of choice for OSA is Continuous Positive Airway Pressure (CPAP). CPAP acts as a positive airway splint, delivering a fixed or auto adjusted positive pressure to the upper airway via a tube and mask. The modified device to be assessed in this study will act in a similar way to the existing device, VPAP Auto, but utilizes an improved algorithm which should maintain or enhance the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Patients who are on CPAP therapy in AUTOSET mode for no less than 6 months
* Patients who are using ResMed masks

Exclusion Criteria:

* Patients who are unable to provide written informed consent
* Patients who are unable to comprehend written and spoken English
* Patients who are using Bilevel PAP
* Patients who are pregnant
* Patients who are suffering any of the following:

  * Acute respiratory infection
  * Acute sinusitis, otitis media or perforated eardrum
  * Pneumothorax or pneumomediastinum
  * Recent history of severe epistaxis requiring medical attention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05-11 (Actual); Primary Completion 2009-06-15 (Actual); Study Completion 2009-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed/The University of New South Wales
Locations (1):
- Centre for Healthy Sleep, Bella Vista, New South Wales, Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Autoset (Nexus Flow Generator): AutoSet algorithms measure breathing patterns and respond to increase or decresase pressures to overcome obstructive sleep apnea. The modified AutoSet algorithm contains software updates to better measure and respond to sleep apnea. Participants used this device for one night, followed by the standard AutoSet, in a randomised order
- VPAP Flow Generator 25: Existing AutoSet algorithm for the treatment of obstructive sleep apnea. Participants used this device for one night, followed by the modified AutoSet algorithm, in a randomised order
Period: Overall Study
Arm/Group | Modified Autoset (Nexus Flow Generator) | VPAP Flow Generator 25
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This was a cross-over study, therefore all participants were assigned to both interventions, for one night each, in a randomised order
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Primary Outcome: Apnoea-Hypopnoea Index (AHI)
Description: The number of apneas and hypopnoeas per hour of sleep measured on Nexus Auto & VPAP Auto 25
Time Frame: One Night On Each Arm, approximately 8 hours each night
Population: Participants included in the study were those who were on CPAP therapy for no less than 6 months and were on auto adjustment mode.
Measure: Mean (Standard Deviation); unit: Events/Hour
Groups:
- Nexus Flow Generator: Participants were randomised to Nexus Flow Generator with modified auto set algorithm group for one night.
- VPAP Flow Generator 25: Participants were randomised to VPAP Flow Generator Auto 25 with A10 algorithm group for one night.
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
Number analyzed (Participants) | 20 | 20
Events/Hour | 1.69 (2.37) | 1.73 (1.58)

2. Primary Outcome: Oxygen Desaturation Index
Description: Number of oxygen desaturations per hour of sleep
Time Frame: One Night On Each Arm, approximately 8 hours each night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Events/Hour
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
Number analyzed (Participants) | 20 | 20
Events/Hour | 1.95 (2.33) | 1.68 (1.35)

3. Secondary Outcome: Comfort of Breathing
Description: Participant's Comfort Rating in one question: How comfortable/uncomfortable was the CPAP device to breathe on? Ratings from 0 (very uncomfortable) to 10 (very comfortable) on a Likert Scale
Time Frame: One Night On Each Arm, approximately 8 hours each night
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a Scale
Groups:
- Nexus Flow Generator: Participants were randomised for Nexus Flow Generator group for one night.
  Nexus Flow Generator: The modified device to be assessed in this study will act in a similar way to the existing device, VPAP Auto, but utilises an improved algorithm which should maintain or enhance the effectiveness of the treatment.
- VPAP Flow Generator 25: Participants were randomised for VPAP Flow Generator 25 group for one night.
  VPAP Flow Generator 25: Exiting VPAP Auto 25 Flow Generator with A10 Algorithm
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
Number analyzed (Participants) | 20 | 20
Scores on a Scale | 8.0 [5 to 10] | 7.0 [7 to 10]

4. Secondary Outcome: Satisfaction of Treatment
Description: Participant's treatment satisfaction in one question: How much did the CPAP disturb your sleep last night? Rating from 0 (a lot) to 10 (not at all) on a Likert Scale
Time Frame: One Night On Each Arm, approximately 8 hours each night
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
Number analyzed (Participants) | 20 | 20
Scores on a scale | 9.5 [5 to 10] | 8.0 [3 to 10]

5. Secondary Outcome: Refreshed Feel
Description: Participants rated 0 (not refreshed at all) to 10 (very refreshed) on Likert Scale on one question: How refreshed did you feel this morning?
Time Frame: One Night On Each Arm, approximately 8 hours each night
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
Number analyzed (Participants) | 20 | 20
Scores on a scale | 9.0 [6 to 10] | 8.0 [5 to 10]

ADVERSE EVENTS:
Time Frame: 2 consecutive nights
Groups:
- Nexus Flow Generator: Modified AutoSet for the treatment of OSA. Participants used this device while sleeping for one night. No Adverse Events were reported during the trial
- VPAP Flow Generator 25: Standard AutoSet for the treatment of OSA. Participants used this device while sleeping for one night. No adverse events were reported during the trial
Arm/Group | Nexus Flow Generator | VPAP Flow Generator 25
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes